CLINICAL TRIAL: NCT06049082
Title: A Phase 1 Study of Inhaled KB408 for the Treatment of Alpha-1 Antitrypsin Deficiency
Brief Title: A Study of KB408 for the Treatment of Alpha-1 Antitrypsin Deficiency
Acronym: Serpentine-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB408-01
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Low dose KB408 (Experimental): Single dose of KB408 (low dose)
  Interventions: Drug: KB408 (Nebulization)
- Cohort 2: Mid dose KB408 (Experimental): Single dose of KB408 (mid dose)
  Interventions: Drug: KB408 (Nebulization)
- Cohort 3: High dose KB408 (Experimental): Single dose of KB408 (high dose)
  Interventions: Drug: KB408 (Nebulization)
- Cohort 2b: Mid dose KB408 (Experimental): Multiple doses of KB408 (mid dose)
  Interventions: Drug: KB408 (Nebulization)

INTERVENTIONS:
Drug: KB408 (Nebulization) — Nebulized solution of KB408, a replication-defective HSV-1 vector expressing full length human SERPINA1

SUMMARY:
The Sponsor is developing KB408, a replication-defective, non-integrating herpes simplex virus type 1 (HSV-1)-derived vector engineered to deliver functional full-length human SERPINA1 to the airways of people with alpha-1 antitrypsin deficiency (AATD) via nebulization. This study is designed to evaluate safety and pharmacodynamics of KB408 in adults with AATD with a PI*ZZ or PI*ZNull genotype. Three planned dose levels of KB408 will be evaluated in single dose escalation cohorts. Repeat dosing will be evaluated at the mid dose level. Subjects taking intravenous AAT augmentation therapy are not required to wash out from IV AAT in the low and mid dose cohorts. In the repeat dose and the high dose cohorts, subjects must wash out from IV AAT for at least 10 days, as applicable.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legally authorized representative must have read, understood, and signed an Institutional Review Board (IRB) approved Informed Consent Form and must be willing and able to comply with study procedures and instructions.
2. Subject is aged ≥18 to ≤70 years, at the time of informed consent.
3. Subject has a genetically confirmed diagnosis of AATD with a PI*ZZ or PI*ZNull genotype.
4. Cohort 2b and Cohort 3: Subjects receiving AAT augmentation therapy must be willing to washout for at least 10 days prior to Screening and be willing to remain off augmentation therapy for the duration of the study.
5. Cohort 2b and Cohort 3: Serum AAT level <11 μM at Screening.
6. Willing to remain on a stable regimen of treatment during the study.
7. Resting oxygen saturation ≥92% on room air at Screening.
8. Clinically stable and in good general health, except for AATD, as determined by the Investigator.

Exclusion Criteria:

1. Pulmonary function test with percent predicted forced expired volume in 1 second (ppFEV1) after inhalation of a bronchodilator is <40% at Screening.
2. Diffusing capacity of the lungs for carbon monoxide (DLCO) <30 percent predicted (historical DLCO within 2 years prior to Screening without any intervening change in clinical status since the measurement was taken, or as measured at Screening).
3. Known ongoing or history of clinically significant pulmonary impairment other than AATD.
4. A pulmonary exacerbation within six weeks (42 days) of first dose.
5. Initiation of any new chronic therapy or any change in ongoing therapy routine within 28 days of first dose.
6. Participation in another interventional clinical study or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, of first dose. Previous treatment with a genetic therapy for AATD, where the investigational product was demonstrated to be non-efficacious, is not exclusionary.
7. History of or listed for solid organ transplantation or has undergone major lung surgery (e.g., lobectomy) within 6 months of first dose.
8. Any clinical condition or illness (including a history or current evidence of substance abuse or dependence) that, in the opinion of the Investigator, would impact a subject's ability to complete all study-related procedures and/or poses an additional risk to the assessment of safety of KB408.
9. An active oral herpes infection 30 days prior to the first dose.
10. Clinically significant hepatic dysfunction defined as any one of the following:

    1. AST and ALT ≥3× upper limit of normal (ULN) at Screening
    2. Total bilirubin ≥2× ULN at Screening (unless associated with Gilbert's syndrome)
    3. Evidence of liver cirrhosis with clinical manifestations of portal hypertension (e.g., ascites, encephalopathy, variceal hemorrhage)
11. History of cigarette smoking or any other tobacco use, or use of e-cigarettes or other recreational inhalant, within 6 months of Screening.
12. Unwilling to refrain from smoking, e-cigarette use, or vaping throughout the duration of the study.
13. A positive urine cotinine result that is consistent with active smoking at Screening. (A positive cotinine test due to nicotine replacement therapy for the purpose of smoking cessation, as attested by the Investigator, is allowed.)
14. Abnormal hematology or chemistry testing at Screening as defined below, or any other clinically significant abnormalities that the Investigator believes may interfere with the assessment of safety of the study treatment.

    * Platelet count <100×10^9/L
    * Hemoglobin <9 g/dL
    * White blood cell count <3 or >15×10^9/L
    * Sodium <130 or >150 mmol/L
    * Potassium <3 or >5.5 mmol/L
    * Carbon dioxide <16 mmol/L
    * Creatinine >2 mg/dL
15. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol, in the opinion of the Investigator.
16. Females who are pregnant or nursing.
17. Subject who is unwilling to comply with contraception requirements per protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of KB408 based upon assessment of adverse events (frequency, severity, relatedness), and changes from baseline in vital signs, ECG, spirometry, and clinical laboratory test results | 2 months (Cohorts 1, 2, 3); 3 months (Cohort 2b)
  Number of subjects with treatment related adverse events as assessed by NCI-CTCAE v5

SECONDARY OUTCOMES:
To assess the effect of KB408 on serum alpha-1 antitrypsin (AAT) concentration | 2 months (Cohorts 1, 2, 3); 3 months (Cohort 2b)
  Change from baseline in serum AAT levels
To assess the effect of KB408 on plasma neutrophil elastase (NE) concentration | 2 months (Cohorts 1, 2, 3); 3 months (Cohort 2b)
  Change from baseline in plasma NE levels
To evaluate the effect of KB408 on AAT concentration in the lung | 2 months (Cohorts 1, 2, 3); 3 months (Cohort 2b)
  Change from baseline in AAT levels in bronchoalveolar lavage fluid
To evaluate the effect of KB408 on NE concentration in the lung | 2 months (Cohorts 1, 2, 3); 3 months (Cohort 2b)
  Change from baseline in NE levels in bronchoalveolar lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: David Sweet, MD, PhD, Study Director — Director of Clinical Development
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Gainesville, Florida
  - Medical University of South Carolina, Charleston, South Carolina
  - Renovatio Clinical, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No